CLINICAL TRIAL: NCT03352011
Title: Primary Care Brief Mindfulness Training for Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse VA Medical Center (U.S. Federal Agency)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Kyle Possemato, Associate Director for Research, Center for Integrated Healthcare, Syracuse VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1147099-1; 5R34AT009678-02 (NIH)
Record Dates: First submitted 2017-11-14; First posted 2017-11-24 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Care Brief Mindfulness Training (Experimental): group-based mindfulness training
  Interventions: Behavioral: Primary Care Brief Mindfulness Training
- PTSD Psychoeducational Class (Active Comparator): group-based psychoeducation class
  Interventions: Behavioral: PTSD Psychoeducational Class

INTERVENTIONS:
Behavioral: Primary Care Brief Mindfulness Training — Primary Care Brief Mindfulness Training consists of four 90-minute group classes that teach sitting meditation, body scan, moving meditation, gentle yoga, and group discussion on topics such as non-judging, patience, trust, non-striving, acceptance, and letting go.
  Arms: Primary Care Brief Mindfulness Training
Behavioral: PTSD Psychoeducational Class — The PTSD Psychoeducational Class is designed to provide a supportive environment for learning about PTSD-related issues and to help Veterans determine what recovery strategies will be most helpful for them. Session themes include "Civilian Readjustment and PTSD," "Trust, Safety, and Healing" and "Treatment Strategies."
  Arms: PTSD Psychoeducational Class

SUMMARY:
The proposed study supports a line of research that seeks to improve the health of military veterans with post-traumatic stress disorder (PTSD) by teaching them mindfulness skills. The proposed study first gathers Veteran's Affairs mental health provider and peer support specialist feedback to adapt a brief mindfulness intervention and then investigates the feasibility of testing this intervention in a small randomized clinical trial. The study targets primary care patients with PTSD who may be reluctant to engage in other mental health treatments and provides them with mindfulness training to reduce PTSD symptoms, improve psychosocial functioning and increase hope for recovery.

DETAILED DESCRIPTION:
Posttraumatic Stress Disorder (PTSD) is highly prevalent in Veterans Affairs (VA) primary care patients (~11.5%) and is associated with significant functional impairment, compromised health, and economic costs. While effective psychotherapies for PTSD are available in VA specialty mental health care settings, primary care patients do not routinely engage in or complete these specialty services. Therefore, alternative delivery models are needed. This proposal integrates two lines of research: mindfulness training and peer support services to test a low-stigma intervention in primary care: Primary Care Based Mindfulness Training (PCBMT). Brief mindfulness training focuses on skill acquisition to help patients manage distress and can serve as a gateway to more intensive treatments for Veterans who are not yet willing to discuss their trauma histories. Peer support specialists help shift treatment away from the medical model focused on symptom reduction to a recovery model focused on leading a meaningful, purposeful life, with or without ongoing illness.

This proposal aims to refine our existing PCBMT to be co-delivered by VA mental health providers and peers and then test important aspects of feasibility to prepare for a future full-scale pragmatic clinical trial. First, VA providers and peers will participate in PCBMT led by study investigators who are certified Mindfulness Based Stress Reduction (MBSR) instructors. Next, study staff will gather feedback from the trained providers and peers for further adaptation and implementation. After this, providers and peers interested in being trained as PCBMT interventionists will be trained by study investigators. Finally, a pilot RCT will be conducted. Both treatments conditions will consist of four, 90-minute group sessions co-facilitated by a VA provider and Veteran peer.

The long-term goal of this research is to improve clinical and personal recovery outcomes for Veterans with PTSD. Our immediate goals are to refine PCBMT based on Veteran, provider, and peer feedback then test the methods needed to conduct a future full-scale RCT, in accordance with the following aims:

1. Gather VA mental health provider (n=5) and peer (n=5) feedback to refine PCBMT to a) ensure successful implementation in the VA setting (including creation of a provider manual and standardized provider/peer training curriculum) and b) maximize Veteran skill development to aid in future participation of evidence-based treatment for PTSD.
2. Assess the feasibility of conducting a pilot RCT (N=60) comparing PCBMT to a PTSD psychoeducation group on a) rates of recruitment and study retention, b) participant adherence and retention in treatment, provider and peer treatment fidelity, c) participant acceptability (satisfaction, perceived helpfulness) in PCBMT and control condition, and d) measuring outcomes of interest for the future larger trial including: PTSD severity, psychosocial functioning, recovery orientation, active engagement in mental health care.

ELIGIBILITY:
Inclusion Criteria:

1. enrolled in services at the Syracuse or Canandaigua VAMC and
2. report significant PTSD symptoms (qualifying criterion A traumatic event plus at least a 31 on the PCL-5).

Exclusion Criteria:

1. gross cognitive impairment (>16 on the Blessed OMC),
2. suicide attempt or desire to commit suicide in the last month (as measured by P4 screener).
3. have received psychotherapy or change in psychiatric medication outside of VHA primary care in the last 2 months.
4. voice a preference to be directly referred to specialty mental health care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Possemato, Ph.D., Principal Investigator — VA Center for Intergrated Healthcare
Locations (1):
- Syracuse Veterans Affairs Medical Center, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Possemato K, Bergen-Cico D, Buckheit K, Ramon A, McKenzie S, Smith AR, Wade M, Beehler GP, Pigeon WR. Randomized Clinical Trial of Brief Primary Care-Based Mindfulness Training Versus a Psychoeducational Group for Veterans With Posttraumatic Stress Disorder. J Clin Psychiatry. 2022 Dec 28;84(1):22m14510. doi: 10.4088/JCP.22m14510. PMID 36576365

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Care Brief Mindfulness Training | PTSD Psychoeducational Class
Started | 28 | 27
Completed | 21 | 20
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Care Brief Mindfulness Training | PTSD Psychoeducational Class | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 12 | 11 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 24 | 24 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 27 | 25 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 26 | 21 | 47
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Assessment Retention Assessment Retention
Description: rate of participants who complete all assessment time points
Time Frame: enrollment to 24 week follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Care Brief Mindfulness Training | PTSD Psychoeducational Class
Number analyzed (Participants) | 28 | 27
Participants | 24 | 25

2. Primary Outcome: Intervention Retention
Description: rate of participants who complete assigned intervention
Time Frame: enrollment to 24 week follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Care Brief Mindfulness Training | PTSD Psychoeducational Class
Number analyzed (Participants) | 28 | 27
Participants | 21 | 20

3. Primary Outcome: Primary Care Brief Mindfulness Fidelity Assessment
Description: Number of essential components of the Primary Care Brief Mindfulness Training curriculum delivered across all 5 cohorts of PCBMT. Number of essential components 0-90. Higher scores indicate more components delivered and better fidelity.
Time Frame: enrollment to 8 week follow-up
Population: Data were not collected for the "PTSD Psychoeducational Class Arm/ Group"
Measure: Number; unit: number of essential components delivered
Arm/Group | Primary Care Brief Mindfulness Training | PTSD Psychoeducational Class
Number analyzed (Participants) | 28 | 0
number of essential components delivered | 85 |

4. Primary Outcome: Client Satisfaction Scale
Description: measured by the Client Satisfaction Questionnaire, scale range 1-32 with 32 indicating highest satisfaction.
Time Frame: 8 week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Primary Care Brief Mindfulness Training | PTSD Psychoeducational Class
Number analyzed (Participants) | 27 | 25
units on a scale | 19.07 (1.174) | 19.36 (1.287)

5. Secondary Outcome: Post-traumatic Stress Checklist for DSM-5
Description: PTSD Checklist-5. Scale range 0-63 with 63 indicating highest PTSD severity.
Time Frame: 24 week follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Primary Care Brief Mindfulness Training | PTSD Psychoeducational Class
Number analyzed (Participants) | 24 | 25
score on a scale | 32.99 (3.27) | 40.89 (3.29)

6. Secondary Outcome: Recovery Orientation Scale- 24
Description: Recovery Orientation Scale-24 measuring recovery from mental health concerns. Range 24-120, with 120 indicating the greatest amount of recovery.
Time Frame: 24 week follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Primary Care Brief Mindfulness Training | PTSD Psychoeducational Class
Number analyzed (Participants) | 24 | 25
score on a scale | 89.53 (2.88) | 82.35 (2.90)

7. Secondary Outcome: Patient Health Questionnaire-9,
Description: Patient Health Questionnaire-9, range 0-27, with 27 indicating the greatest amount of depression.
Time Frame: 24 week follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Primary Care Brief Mindfulness Training | PTSD Psychoeducational Class
Number analyzed (Participants) | 24 | 25
score on a scale | 9.12 (1.21) | 12.98 (1.21)

8. Secondary Outcome: Self Compassion Scale- Short Form
Description: Self Compassion Scale- Short Form, range 0-60, with 60 indicating the greatest amount of self compassion.
Time Frame: 8 week post-treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Primary Care Brief Mindfulness Training | PTSD Psychoeducational Class
Number analyzed (Participants) | 27 | 25
score on a scale | 32.38 (1.40) | 34.34 (1.98)

9. Secondary Outcome: Health Promoting Lifestyle Profile II: Health Responsibility Subscale
Description: Health Promoting Lifestyle Profile II: Health Responsibility. Subscale ranges from 9-36, with 36 indicating the most health responsibility.
Time Frame: 24 week follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Primary Care Brief Mindfulness Training | PTSD Psychoeducational Class
Number analyzed (Participants) | 24 | 25
score on a scale | 24.80 (1.00) | 21.40 (1.00)

ADVERSE EVENTS:
Time Frame: enrollment to 24 weeks
Arm/Group | Primary Care Brief Mindfulness Training | PTSD Psychoeducational Class
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25
Serious Adverse Events (participants affected / at risk) | 3/27 | 4/25
Other Adverse Events (participants affected / at risk) | 0/27 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Care Brief Mindfulness Training (N=27) | PTSD Psychoeducational Class (N=25)
ER visit or hospitalization unrelated to study interventions (General disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT03352011/Prot_SAP_000.pdf